CLINICAL TRIAL: NCT05596357
Title: Observational Study of the Benefits of Complex Abdominal Wall Repairs on Quality of Life , Digestive and Sexual Functions.
Brief Title: Incisional heRnia dIgestion Sexuality
Acronym: IRIS
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A01003-38
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaires — The patient must answer questionnaires before and after reconstructive surgery

SUMMARY:
After an operation on the abdomen, some patients present with an incisional hernia(incisional hernia) which causes a permanent exteriorization of the vicera. This situation is at the origin of postural problems. Surgery which consists both of reducing pain and correcting the functional limitation and aesthetic damage helps restore normal anatomy and improve muscle tension of the wall, restore the musculoskeletal balance of the trunk and thus the cardio-respiratory and motor functions of patients. The resulting benefits on quality of life and reduction of chronic pain have been demonstrated by several studies. This study tends to better understand the functional and sexual prejudices linked to these parietal pathologies by passing questionnaires to the operated patients

DETAILED DESCRIPTION:
Almost 20% of patients operated on the abdomen will present with an incisional hernia and each year in France, more than 50,000 patients are operated on for an eventration with placement of a parietal mesh.

These incisional hernia, corresponding to the permanent exteriorization of the abdominal viscera contained in a peritoneal sac through a scar muscle defect in the abdominal wall, are responsible for major anatomical and physiological alterations affecting the respiratory, cardiovascular and musculoskeletal systems.

Sometimes the hernia sac is so large that the viscera have lost their place in the abdomen . The presence of a large protrusion of the anterior abdomen alters the patient's center of gravity, affecting his ambulation and posture

Thus, surgical repair of the abdomen, indicated to correct chronic pain, functional limitation and cosmetic damage related to incisional hernia, helps restore normal anatomy and improve muscle tension of the wall, restore the musculoskeletal balance of the trunk and thus the cardio-respiratory and motor functions of the patients. The consequent benefits on the quality of life and the reduction of chronic pain have been demonstrated by several studies, including a randomized trial [Rogmark, but certain aspects of the functional limitations linked to the presence of an eventration have never been studied (not published), as well as their specific impact on quality of life.

In fact, the daily experience of the management of these pathologies suggests that most patients with an abdominal wall problem, on the one hand, evoke difficulties to exonerate (abdominal pushing efforts are rendered ineffective due to the leakage of abdominal pressure in the incisional hernia sac, sometimes forcing patients to contain their stomachs by manual maneuvers or to wear an abdominal belt) and on the other hand difficulty having sexual intercourse (gene linked to the protrusion of abdomen, impaired body image and self-esteem).

Thus, a better knowledge of the actual digestive and sexual functional damage linked to these parietal pathologies, will make it possible to optimize the care of patients who will be better informed about their disease and the benefits they can expect from parietal repair (ease of having a bowel movement, improvement of sex life, benefits on quality of life).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 79
* No opposition to research
* Planned surgery to cure a hernia or complex anterior eventration of the abdomen by laparotomy or laparoscopy
* Mastery of the French language sufficient to answer questionnaires

  * Registration in a national health care system

Exclusion Criteria:

* Emergency surgery
* ASA (American Society of Anesthesiologists) score> 3 during the preoperative consultation
* Current pregnancy or breastfeeding
* Patient under guardianship or curatorship
* Patient under AME (State Medical Aid)

Ages: 18 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients operated on on the abdomen will present with an eventration (incisional hernia)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Symtoms of constipation --> Patient Assessment of Constipation Symptoms (PAC-SYM) | 25 months
  Analyze changes in symptoms related to constipation before (1 month) and after surgical operation (M3, M12 and M24)

SECONDARY OUTCOMES:
Quality of life related to constipation -->Patient Assessment of Constipation Quality of Life questionnaire (PAC-QOL) | 25 months
  Assessment of qualitiy of life related to constipation before (1 month) and after surgical operation (M3, M12 and M 24)
Quality of life related to digestive function--> Gastrointestinal Quality of Life index (GIQLI) | 25 months
  Assessment of qualitiy of life related to digestive function before (1 month) and after surgical operation (M3, M12 and M 24)

OTHER OUTCOMES:
Analysis of sexual function -->Femal Sexual Function Index (FSFI) and Male Sexual Health Questionnaire (MHSQ). | 25 months
  Analyze changes in sexual function before (1 month) and after surgical operation (M3 M12, M24)
Changes in quality of life analysis --> Medical Outcome Study Short Form 12 (SF12), | 25 months
  Analyze changes in quality of life before (1 month) and after surgical operation (M3 M12, M24)
Clinical recurrence | 36 months
  Assessment of clinical recurrence M1, M3, M6, M12, M24, M36 after surgical operation
Radiological recurrence | 24 months
  Assessment of radiological recurrence at M24 after surgical operation
Death | 36 months
  Assessment of the mortality up to M36 after surgical operation
Pain analysis--> Visual Analog Scale (VAS) | 36 months
  Analyze postoperative pain: M1, M3, M6, M12, M24 and M36
Morbidity --> Sepsis on mesh, hematoma, seroma, reoperation for complication, removal of the parietal mesh. | 1 month
  Assessment of morbidity after surgical operation

CONTACTS AND LOCATIONS:
Locations (1):
- David Moszkowicz, Colombes, Île-de-France Region, France